CLINICAL TRIAL: NCT02737943
Title: Randomized Single-center, Single-blind, Two-arm Parallel Group Trial of Using MEBO™ Dressing Versus Standard Care at Zagazig University Hospital in the Management of Donor and Recipient Sites of Split-thickness Skin Graft
Brief Title: Effect of Mebo Dressing Versus Standard Care on Managing Donor and Recipient Sites of Split-thickness Skin Graft
Acronym: EMD-SCZ-SGS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohammad Alsabbahi, DR, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2579
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Burns
Keywords: Skin graft; Burn; MEBO; Wound dressing; Wound care; Raw Area
MeSH Terms: conditions — Burns | interventions — moist exposed burn ointment; Anti-Bacterial Agents; Analgesics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1 Mebo (Experimental): 20 : receiving Moist Exposed Burn Ointment (MEBO) at sites of donor graft and recipient at time of operation and in dressing
  Interventions: Drug: Moist Exposed Burn Ointment (MEBO)
- Arm2 Placebo (Placebo Comparator): 20 : receiving Standard cream Zagazig University Hospital (Antibiotics & analgesics)
  Interventions: Drug: Zagazig

INTERVENTIONS:
Drug: Moist Exposed Burn Ointment (MEBO) — is a registered USA patented formulation since 1995. MEBO is pure herbal, natural in origin, containing beta-sitosterol phellodendron amurense, scutellaria baicalensis, coptis chinensis, pheretima aspergillum, Beeswax and sesame oil. 15, 19 The pharmacological effects are attributable to: beta-sitosterol, isolated from phellodendron amurense, flavonoids mainly baicalin isolated from scutellaria baicalensis, alkaloids mainly berberine, isolated from coptis chinensis, Beeswax and sesame oil.
  Other Names: MEBO cream
  Arms: Arm1 Mebo
Drug: Zagazig — Standard care is an antibiotic ointment in combination of analgesic for relief of pain.
  Other Names: Antibiotic & Analgesic
  Arms: Arm2 Placebo

SUMMARY:
40 Egyptian Cases with split-thickness skin graft receiving treatment at Zagazig University Hospitals. Study Duration:6 Months .Description of Agent or Moist Exposed Burn Ointment (MEBO).

Intervention:

Objectives: Primary: to determine the efficacy of MEBO versus standard care in improving the healing speed and re-epithelization process of skin graft donor and recipient sites. Secondary to determine the efficacy of MEBO in decreasing recovery time, rate of infections, rate of complications, total treatment costs and its effect on improving pain alleviation.

Description of Study Design: Arm 1 20 MEBO at sites of donor graft and recipient at time of operation and in dressing Arm 2 20 Standard cream Zagazig University Hospital (Antibiotics & analgesics) Estimated Time to Complete 5 months

DETAILED DESCRIPTION:
Background Information.

Skin grafting is a frequently used technique for covering skin defects in cases of row area. The technique evolved from use in the back alleys of India in pre-Christian times to become one of the most valuable clinical tools in modern surgery. There are several techniques for caring for the skin graft site to assure an adequate graft and prompt as well as wound healing.

The use of the split-thickness skin graft (STSG) as reconstructive technique is very common nowadays but this technique is usually a source of pain and discomfort for the patients and may cause significant morbidity and result in hypertrophic or even keloid scarring. The wound heals by a process of re-epithelialization which results in an epithelial cover usually within 7-14 days. The aim of graft management is to maintain an environment that promotes optimal healing and prevents morbidity, which can include pain and infection and ultimately delayed healing.

The dressing of donor and recipient sites which provides a protective barrier should be easy to apply, promote rapid re-epithelialization, and be pain free, infection free, and relatively inexpensive.

MEBO have been proved to have anti-inflammatory and anti-microbial effect due to the presence of - β sitosterol and berberine respectively. Many studies have reported that MEBO provides suitable moist environment needed for burn wounds for optimal healing and re-epithelialization without the need for wound closure by dressing. Also some studies have proved the efficacy of MEBO in secondary healing of partial thickness wounds, such as split thickness skin graft sites, with improved cosmetic results and better scar quality.

In cases of raw area, donor and recipient sites have been traditionally dressed with low-adherent wound contact paraffin gauze or antibiotic-impregnated tulle gras and covered by a secondary dressing made of gauze and absorbent padding.

These dressings are relatively inexpensive. However, during the peri-operative period, patients complain more often of discomfort or pain at the donor area than at the graft site itself besides, the poor cosmetic appearance of donor sites after healing is not readily accepted.

Because the basic pathology of burns closely mimics many aspects of skin graft donor sites, researchers are investigating using MEBO at donor and recipient sites.

Potential Risks

Due its pure and natural origin, MEBO have been reported to have no side effect or potential risks except rare cases of allergy and hypersensitivity.

Known Potential Benefits

MEBO has been proved to have a positive effect on improving healing process with rapid re-epithelialization. According to a recent study, the burn areas and graft sites were markedly less hyperemic and less pigmented and the final cosmetic appearance and patient satisfaction were also higher by using MEBO. The cases who used MEBO had better scar assessment and lower pain scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be managed using split-thickness skin graft.
2. Donor skin grafts are harvested from a site in the thigh (a minimum of 5 x 5-cm total area).
3. Intention for treatment at Zagazig University.
4. Age between 2 & 60 years.
5. An approved informed consent and authorization permitting release of personal health information must be signed by patient or guardian.
6. Compliance with treatment for 3 weeks.
7. Patients of childbearing age must have a negative pregnancy test.

Exclusion Criteria:

1. Chemical or electrical burns.
2. Patient with concomitant injury of head trauma, inhalation injury, or bone fracture.
3. Pregnant or breast-feeding female.
4. Known or suspected allergies to any of the components of MEBO.
5. Suspicion or presence of active systemic or local cancer or tumor of any kind.
6. Any immune deficiency disorder.
7. Suspected alcohol or drug abuse.
8. Participation in another investigational drug study within 30 days prior to treatment start.
9. If the donor site is less than 5 x 5-cm total area.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Wound Healing Assessment | 1 month
  Standardized digital photographs will be taken of each site at the time of wound inspection, visit 1 and visit 2 then a plastic surgeon and a plastic resident will assessed the healing process blindly. These observers independently will rate the extent of re -epithelialization in each image as none, less than 50%, more than 50% but not complete, or complete. A numeric score was given to each rating as follows:
  No re epithelialization=0, less than 50%=1, more than 50%=2, and complete=3. Hence, a higher score indicated a greater estimated extent of re -epithelialization.

SECONDARY OUTCOMES:
Recovery Time | 1 month
  Time from randomization till primary healing of 75% raw area surface are (BSA) and complete secondary healing of skin graft.
Rate of Infections | 2 weeks
  Clinical assessment to detect early signs of infections and Culture for further investigations.
Pain Assessment | 2 weeks
  Visual analogue scale (VAS) of pain (0-10); 0 is the minimum and 10 is the maximum Recording type and dose of administrated analgesics.
Total Treatment Costs | 1 month
  Costs including (administrated medications, examinations costs, follow up visits after discharge).
Rate of Complications | 1 week
  Rates of allergy, infection and bleeding rate
Quality of Life | 1 month
  Health related quality of life (HRQL) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad H Abdel-All, Professor, Study Director — Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Alsharkia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atiyeh BS, Dham R, Kadry M, Abdallah AF, Al-Oteify M, Fathi O, Samir A. Benefit-cost analysis of moist exposed burn ointment. Burns. 2002 Nov;28(7):659-63. doi: 10.1016/s0305-4179(02)00075-x. PMID 12417161
- [Background] Mabrouk A, Boughdadi NS, Helal HA, Zaki BM, Maher A. Moist occlusive dressing (Aquacel((R)) Ag) versus moist open dressing (MEBO((R))) in the management of partial-thickness facial burns: a comparative study in Ain Shams University. Burns. 2012 May;38(3):396-403. doi: 10.1016/j.burns.2011.09.022. Epub 2011 Nov 17. PMID 22100189
- [Background] Carayanni VJ, Tsati EG, Spyropoulou GC, Antonopoulou FN, Ioannovich JD. Comparing oil based ointment versus standard practice for the treatment of moderate burns in Greece: a trial based cost effectiveness evaluation. BMC Complement Altern Med. 2011 Dec 1;11:122. doi: 10.1186/1472-6882-11-122. PMID 22132709
- [Background] Atiyeh BS, Ghanimeh G, Kaddoura IL, Ioannovich J, Al-Amm CA. Split-thickness skin graft donor site dressing: preliminary results of a controlled, clinical comparative study of MEBO and Sofra-Tulle. Ann Plast Surg. 2001 Jan;46(1):87-8. doi: 10.1097/00000637-200101000-00023. No abstract available. PMID 11192048
- [Background] Spear M, Bailey A. Treatment of skin graft donor sites with a unique transparent absorbent acrylic dressing. Plast Surg Nurs. 2009 Oct-Dec;29(4):194-200; quiz 201-2. doi: 10.1097/PSN.0b013e3181c4cdd9. PMID 20029295
- [Background] Weber RS, Hankins P, Limitone E, Callender D, Frankenthaler RM, Wolf P, Goepfert H. Split-thickness skin graft donor site management. A randomized prospective trial comparing a hydrophilic polyurethane absorbent foam dressing with a petrolatum gauze dressing. Arch Otolaryngol Head Neck Surg. 1995 Oct;121(10):1145-9. doi: 10.1001/archotol.1995.01890100055009. PMID 7546582
- [Background] Wiechula R. The use of moist wound-healing dressings in the management of split-thickness skin graft donor sites: a systematic review. Int J Nurs Pract. 2003 Apr;9(2):S9-17. doi: 10.1046/j.1322-7114.2003.00417.x. PMID 12694482
- [Background] Innes ME, Umraw N, Fish JS, Gomez M, Cartotto RC. The use of silver coated dressings on donor site wounds: a prospective, controlled matched pair study. Burns. 2001 Sep;27(6):621-7. doi: 10.1016/s0305-4179(01)00015-8. PMID 11525858
- [Background] Barnea Y, Amir A, Leshem D, Zaretski A, Weiss J, Shafir R, Gur E. Clinical comparative study of aquacel and paraffin gauze dressing for split-skin donor site treatment. Ann Plast Surg. 2004 Aug;53(2):132-6. doi: 10.1097/01.sap.0000112349.42549.b3. PMID 15269581
- [Background] Hormbrey E, Pandya A, Giele H. Adhesive retention dressings are more comfortable than alginate dressings on split-skin-graft donor sites. Br J Plast Surg. 2003 Jul;56(5):498-503. doi: 10.1016/s0007-1226(03)00195-4. PMID 12890465
- [Background] Giele H, Tong A, Huddleston S. Adhesive retention dressings are more comfortable than alginate dressings on split skin graft donor sites--a randomised controlled trial. Ann R Coll Surg Engl. 2001 Nov;83(6):431-4. PMID 11777142